#### Statistical Analysis Plan: Mock-up Subject Data Listing

SCB01A for Metastatic Squamous Cell Head and Neck Cancer

# Statistical Analysis Plan: Mock-up Subject Data Listings

Version 3.0, 14DEC2018

**Protocol Number: SCB01A-22** 

An Open-Label, Phase II Study to Evaluate the Efficacy and Safety of SCB01A in Subjects with Recurrent or Metastatic Squamous Cell Head and Neck Cancer Who Have Failed Platinum-Based Treatment

Protocol version: 1.0/19-Dec-2016 Sponsor: SynCore Biotechnology Co., Ltd.

Version 3.0, 14DEC2018 Protocol No.: SCB01A-22 Confidential Page 1 of 8

SynCore Biotechnology Co., Ltd. Prepared by: A2 Healthcare Taiwan Corporation

# 

#### Statistical Analysis Plan: Mock-up Subject Data Listing

SCB01A for Metastatic Squamous Cell Head and Neck Cancer

The Mock-up "PATIENT DATA LISTINGS" is planned according to ICH E3, in which relevant CSR section is 16.2. The words shadowed below are for notifications, or to be revised, or variables/format/footnotes to be included.

All listing will be sorted by (1) Eligibility {Eligible subjects, Screen failures} (2) Subject ID (3) Visit No. (4) Item No.

#### Note:

(1) The subject ID is auto generate as Site ID - Screening Number - Stage code and Subject Number (C-SX X-SYY) for eligible subject or as Site ID - Screening Number (C-SXX) for screening failure

**Site ID**.: one-digit number C

| Site ID | Site Name |
|---------|-------------------------------------------------------|
| 1 | Taipei Medical University Hospital (TMUH) |
| 2 | National Cheng Kung University Hospital (NCKUH) |
| 3 | Taipei Veterans General Hospital (TVGH) |
| 4 | Taipei Medical University Shuang Ho Hospital (TMUSHH) |

**Screening number**: two-digit number XX assigned sequentially from 01 for each site

**Stage code**: one-digit number **S** {1 - Stage I, 2 - Stage II}

**Subject number**: two-digit number YY assigned sequentially from 01 for each site

#### (2) DP/AG:

D denotes maximum treatment dose level

12: Level 1 (12 mg/m²) 9: Level 1a (9 mg/m²) 7: Level 1b (7 mg/m²) 18: Level 2 (18 mg/m²) 15: Level 2a (15 mg/m²) 12: Level 2b (12 mg/m²) 24: Level 3 (24 mg/m²) 20: Level 3a (20 mg/m²) 16: Level 3b (16 mg/m²)

P denotes population with value of either one below

I: Intent-to-treat (ITT) population

P: Per-protocol (PP) population, ITT included

A denotes age in Y/O

Age [Y/O] = year of informed consent – year of birth

G denotes gender,

M: male, F: female

(3) Date format: YYYY-MM-DD

(4) For Visit Name, C(c) denotes cycle (c), D(d) denotes day (d)

| Visit No. | Visit Name | Visit<br>Code | Planned Visit Day |
|---|---|---|---|
| 0 | Screening Visit | SV | <b>-28</b> ∼ <b>-1</b> |
| 1.01 | Cycle 1 Day 1 | C1D1 | 1 |
| 1.08 | Cycle 1 Day 8 | C1D8 | 7±1 days after C1D1 |
| 1.15 | Cycle 1 Day 15 | C1D15 | 14±2 days after C1D1 |
| c.01 | Cycle © Day 1 | CcD1 | 21±1 days after Ck1D1<br>k=c-1 |
| c.08 | Cycle © Day 8 | CcD8 | 7±1 days after CcD1 |
| c.15 | Cycle © Day 15, ©=1, 2, 3 only | CcD15 | 14±2 days after CcD1 |

Version 3.0, 14DEC2018 Protocol No.: SCB01A-22 Confidential Page 2 of 8

SynCore Biotechnology Co., Ltd. Prepared by: A2 Healthcare Taiwan Corporation



#### Statistical Analysis Plan: Mock-up Subject Data Listing

SCB01A for Metastatic Squamous Cell Head and Neck Cancer

| Visit No. | Visit Name | Visit<br>Code | Planned Visit Day |
|---|---|---|---|
| | End of Treatment (EOT) / Early Withdrawal (EW) | EOT /<br>EW | EOT: 21±2 days after Ck1D1 or 14±2 days after Ck1D8, k=c-1 EW: after the last treatment dose |
| | Toxicity Follow-Up Visit (TFU) | TFU | 28±3 days after the last treatment dose |
| 99.1 | Follow-Up Visit 1 (FU1) | FU1 | 21±3 after EOT/EW |
| 99.2 | Follow-Up Visit 2 (FU2) | FU2 | 21±3 after FU1-W3 |
| 99.3 | Follow-Up Visit 3 (FU3) | FU3 | 21±3 after FU2-W6 |
| 99. F | Follow-Up Visit F (FUF) | FU[F] | Every 9 weeks ±7 days |
| 66. <u>x</u> x | Unscheduled Visit (UV) | UV | |

 $<sup>\</sup>boxed{c}$ : cycle number where  $\boxed{c} \ge 2$ ,  $\boxed{F}$ : assigned sequentially from 4,  $\boxed{x}$ : assigned sequentially from 01

## (5) For the visit/assessment days and hour (like AE Onset Day), they were derived by formula below

Day (D) = date-first dosing date + 1 if date  $\ge$  1st dosing date, or = date-first dosing date if date < 1st dosing date

Day/Hour = [visit/assessment date/time –  $1^{st}$  dosing date/time + 1], if date  $\ge 1^{st}$  dosing date/time,

Day/Hour = [visit/assessment date/time –  $1^{st}$  dosing date/time], if date  $< 1^{st}$  dosing date/time,

Duration in days/hours = [end date/time – onset date/time + 1] if end date/time is active

Duration in days/hours = [end date/time – onset date/time] if end date/time is inactive

#### (6) Full term for 'Primary System Organ Class' in AE:

| Code | Full Term |
|-------|---------------------------------------------------------------------|
| Blood | Blood and lymphatic system disorders |
| Cardi | Cardiac disorders |
| Conge | Congenital, familial and genetic disorders |
| Ear a | Ear and labyrinth disorders |
| Endoc | Endocrine disorders |
| Eye d | Eye disorders |
| Gastr | Gastrointestinal disorders |
| Gener | General disorders and administration site conditions |
| Hepat | Hepatobiliary disorders |
| Immun | Immune system disorders |
| Infec | Infections and infestations |
| Injur | Injury, poisoning and procedural complications |
| Inves | Investigations |
| Metab | Metabolism and nutrition disorders |
| Muscu | Musculoskeletal and connective tissue disorders |
| Neopl | Neoplasms benign, malignant and unspecified (incl cysts and polyps) |
| Nervo | Nervous system disorders |
| Pregn | Pregnancy, puerperium and perinatal conditions |
| Psych | Psychiatric disorders |
| Renal | Renal and urinary disorders |
| Repro | Reproductive system and breast disorders |
| Respi | Respiratory, thoracic and mediastinal disorders |
| Skin | Skin and subcutaneous tissue disorders |
| Socia | Social circumstances |
| Surgi | Surgical and medical procedures |
| Vascu | Vascular disorders |

#### (7) Full term for Laboratory Measurements:

#### Hematology

| LBSPID | Code | Full Term |
|--------|------|-----------|
| LB01 | RBC | RBC |



### **Statistical Analysis Plan:** Mock-up Subject Data Listing SCB01A for Metastatic Squamous Cell Head and Neck Cancer

| I DCDID | Cada | E11 T |
|---|---|---|
| LBSPID | Code | Full Term |
| LB02 | HGB | Hemoglobin |
| LB03 | HCT | Hematocrit |
| LB04 | PLAT | Platelet |
| LB05 | NEUT | Absolute neutrophil count (ANC) |
| LB06 | MCV | Mean Corpuscular Volume (MCV) |
| LB07 | MCH | Mean Corpuscular Hemoglobin (MCH) |
| LB08 | MCHC | Mean Corpuscular Hemoglobin Concentration (MCHC) |
| LB09 | WBC | WBC |
| LB10 | NEUTLE | Neutrophils |
| LB11 | LYMLE | Lymphocytes |
| LB12 | MONOLE | Monocytes |
| LB13 | EOSLE | Eosinophils |
| LB14 | BASOLE | Basophils |
| Biochemis | trv | |
| LBSPID | Code | Full Term |
| LB15 | BILI | Bilirubin (total) |
| LB16 | ALP | Alkaline Phosphatase |
| LB17 | ALT | Alanine aminotransferase |
| LB17<br>LB18 | AST | Aspartate aminotransferase Aspartate aminotransferase |
| LB19 | GGT | Gamma-glutamyl transferase (GGT) |
| LB19<br>LB20 | ALB | Albumin |
| LB20<br>LB21 | PROT | |
| | | Total protein |
| LB22 | CREAT | Creatinine |
| LB23 | BUN | Blood urea nitrogen (BUN) |
| LB24 | URIAC | Uric Acid |
| LB25 | CK | Creatinine Kinase (Ck) |
| LB26 | TROPONT | Troponin-T |
| LB27 | TROPONI | Troponin-I |
| LB28 | SODIUM | Sodium (Na+) |
| LB29 | K | Potassium (K+) |
| LB30 | CA | Calcium (Ca++) |
| LB31 | CL | Chloride (Cl) |
| LB32 | GLUC | Glucose |
| LB33 | TRIG | Triglycerides (TG) |
| LB34 | AMYLASE | Amylase |
| LB35 | CREATCLR | Creatinine Clearance |
| LB36 | CHOL | Total Cholesterol |
| LB37 | HDL | High-Density Lipoprotein (HDL) |
| LB38 | LDL | Low-Density Lipoprotein (LDL) |
| LB39 | LIPASE | Lipase |
| Coagulatio | | Lipuse |
| LBSPID | Code | Full Term |
| LB40 | PT | Prothrombin Time |
| | | Prothrombin Intl. Normalized Ratio |
| LB41 | INR | Prountomoin inti. Normalized Ratio |
| Urinalysis | G 1 | p tim |
| LBSPID | Code | Full Term |
| LB42 | UPH | pH |
| LB43 | APPEAR | Appearance |
| LB44 | COLOR | Color |
| LB45 | SPGRAV | Specific gravity |
| LB46 | VISC | Viscosity |
| LB47 | TURB | Turbidity |
| LB48 | KETONES | Ketones |
| LB49 | UBILI | Bilirubin |
| I D50 | OCCDI D | Pland |

OCCBLD

LB50

Blood



### **Statistical Analysis Plan:** Mock-up Subject Data Listing SCB01A for Metastatic Squamous Cell Head and Neck Cancer

| LBSPID | Code | Full Term |
|--------|----------|---------------------|
| LB51 | UGLUC | Glucose |
| LB52 | UPROT | Protein |
| LB53 | NITRITE | Nitrite |
| LB54 | UROBIL | Urobilinogen |
| LB55 | LEUKASE | Leukocyte esterases |
| LB56 | BACT | Bacteria |
| LB57 | CASTS | Casts |
| LB58 | CRYSTALS | Crystals |
| LB59 | EPIC | Epithelial Cells |
| LB60 | URBC | RBC |
| LB61 | UWBC | WBC |

- (8) For clinical relevant,
  CS denotes 'abnormal and clinically significant',
  NCS denotes 'abnormal but not clinically significant'

#### (9) General Abbreviations

| Code | Full Term |
|------------|------------------------|
| A, NA, N/A | Not Applicable |
| U, UK, U/K | Unknown |
| O, OG, O/G | Ongoing |
| D, ND, N/D | Not Done |
| M, MS, M/S | Missing |
| MH | Medical History |
| AE | Adverse Event |
| CM | Concomitant Medication |
| INCXX | Inclusion Criterion XX |
| EXCXX | Exclusion Criterion XX |

# ◇ 古輝醫業集團 SynCore Bio

#### Statistical Analysis Plan: Mock-up Subject Data Listing

SCB01A for Metastatic Squamous Cell Head and Neck Cancer

#### **16.2 Patient Data Listings**

#### **16.2.1** Discontinued Subjects

16.2.1.1 Screen Failures

Criteria not met (IE)

16.2.1.2 Study Termination of Eligible Subjects

Domain [DS], including

First Treatment Date/Time,

Last Treatment Date/Time,

End date of treatment phase,

Study Duration (see 14.1.2),

Status (Study Completed or Early Termination),

Reason

16.2.1.3 Inform Consent Date, Visit Dates

#### 16.2.2 Protocol Deviations

- 16.2.2.1 Protocol Deviations Inclusion/Exclusion Subjects
- 16.2.2.2 Protocol Deviations

#### 16.2.3 Eligible Patients Excluded from the Safety/Efficacy Analysis

- 16.2.3.1 Eligible Patients Excluded from Intent-To-Teat (ITT) Population
- 16.2.3.2 Eligible Patients Excluded from Per-protocol (PP) Population
- 16.2.3.3 Eligible Patients Excluded from Pharmacokinetics (PK) Population

#### 16.2.4 Demographic Data and Baseline Characteristics

- 16.2.4.1 Demographic Data
- 16.2.4.2 Smoking Status and Betelnut Consumption
- 16.2.4.3 Head and Neck Squamous Cell Carcinoma (HNSCC) History & Tumor Staging including Disease Duration (see 14.1.4)
- 16.2.4.4 Virology Test and Pregnancy Test
- 16.2.4.5 General Medical History

#### **16.2.5** Medication History and Concomitant Medications

- 16.2.5.1 Cancer Therapy Surgery
- 16.2.5.2 Cancer Therapy Anti-Cancer Medication
- 16.2.5.3 Cancer Therapy Radiotherapy
- 16.2.5.4 Medication History & Concomitant Medications

#### 16.2.6 Study Drug Administration

16.2.6.1 BSA Calculation, SCB01A IV Infusion and Dose Modification

Cycle, Day, Dose Level, BSA  $(m^2) = [Height (cm) \times Body Weight (kg)/3600] \frac{1}{2}$ 

16.2.6.2 BSA Calculation, SCB01A IV Infusion and Dose Modification - Comment / Not Done Reason

16.2.6.3 Study Drug Exposure (See 14.1.6)

# **SynCore**Bio

#### Statistical Analysis Plan: Mock-up Subject Data Listing

SCB01A for Metastatic Squamous Cell Head and Neck Cancer

#### 16.2.7 Efficacy Data

- 16.2.7.1 Radiological Image Assessment Target Lesions
- 16.2.7.2 Radiological Image Assessment Non-Target Lesions
- 16.2.7.3 Radiological Image Assessment Not Done Reason
- 16.2.7.4 Radiological Image Assessment Best Tumor Size Change in Target Lesions
- 16.2.7.5 Tumor Response Assessment

  Including Target Lesions, Non-Target Lesions, Overall Response
- 16.2.7.6 Survival Follow-up
- 16.2.7.7 Cancer Therapy Follow-up
- 16.2.7.8 Overall Efficacy Endpoints

*Including Objective Response (Rate of CR+PR)*,

Date of Death (+ denotes the last survival observation date when death is not observed),

Overall Survival (+ denotes censored at the last survival observation date),

Date of Progression (+ denotes the last tumor assessment date when progression is not observed),

Progression-Free Survival (+ denotes censored at the last tumor assessment date), Best Overall Tumor Response

#### 16.2.8 Adverse Event (AE) and Serious Adverse Event (SAE)

16.2.8.1 Treatment Emergent AEs

Variables: In addition to event description and general AE profiles (onset date, resolution date, severity, relationship to study treatment, action taken to study treatment, seriousness, outcome), the patient data listing will also present the MedDRA(version 19.1) body system and preferred term, onset day, and AE duration [days]

#### Footnote:

- Onset Day = onset date the first treatment dosing date + 1
- AE duration [days]

= resolution date - onset date (while resolved)

=study exit date - onset date (while not resolved, noted with '+')

- 16.2.8.2 Treatment Emergent AEs DLT
- 16.2.8.3 Treatment Emergent AEs Grade ≥3 AEs
- 16.2.8.4 Treatment Emergent AEs Treatment Related AE

Treatment Related is defined as Definitely Related, Probable Related, or Possibly Related

16.2.8.5 Treatment Emergent AEs – Treatment Modified AE

Treatment Modified is defined as Treatment Infusion Interrupted, Treatment Omitted, Dose Reduced, Treatment Discontinued

- 16.2.8.6 Serious Adverse Event
- 16.2.8.7 General Medical History of Subjects with SAE
- 16.2.8.8 Medication History & Concomitant Medications of Subjects with SAE

#### **16.2.9** Laboratory Measurements

- 16.2.9.1 Laboratory Measurements Summary in Standard Unit
- 16.2.9.2 Laboratory Measurements Hematology
- 16.2.9.3 Laboratory Measurements Biochemistry

Version 3.0, 14DEC2018 Confidential SynCore Biotechnology Co., Ltd. Prepared by: A2 Healthcare Taiwan Corporation



### **Statistical Analysis Plan:** Mock-up Subject Data Listing SCB01A for Metastatic Squamous Cell Head and Neck Cancer

| 16.2.9.4 | Laboratory Measurements – Coagulation |
|---|---|
| 16.2.9.5 | Laboratory Measurements – Urinalysis |
| 16.2.9.6<br><b>16.2.10</b> Ot | Laboratory Measurements – Comment and Not Done Reason her Safety Measurements |
| 16.2.10.1 | Vital Signs, Body Weight and ECOG Performance Status |
| 16.2.10.2 | Nerve Conduction Velocity (NCV) |
| 16.2.10.3 | 12-Lead Electrocardiogram (ECG, EKG) |
| 16.2.10.4 | Physical Examination |
| 16.2.10.5 | Physical Abnormalities |
| 16.2.11 Ph | armacokinetic Analysis |
| 16.2.11.1 | Pharmacokinetic Blood Sampling Date/Time |
| 16.2.12 Co | omments |

16.2.12.1 Comments